CLINICAL TRIAL: NCT00481039
Title: Sickle Cell Anemia in an Arab Bedouin Village in the Northern Israel- An Observational Study
Brief Title: Sickle Cell Anemia in an Arab Bedouin Village in the Northern Israel
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dr Koren Ariel, Pediatric Hematology Unit - Ha'Emek Medical Center
Other Study IDs: 5311006.EMC
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Sickle cell thalassemia; Population screening
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Health Records, Personal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients diagnosed as having abnormal hemoglobin like hemoglobin S and thalassemia in a bedouin village
  Interventions: Procedure: Medical history and basic laboratory analysis

INTERVENTIONS:
Procedure: Medical history and basic laboratory analysis — Medical history and basic laboratory analysis

SUMMARY:
Sickle cell anemia and sickle cell thalassemia are frequent diseases among the israeli arab population. The purpose of this study is to assess the clinical characteristics of the patients in one arab village and the laboratory characteristics in the carriers of this gene based in the screening for pregnant women that is carried out in the population of northern Israel.

The results can be useful in order to institute universal screening for sickle cell anemia in northern Israel.

ELIGIBILITY:
Inclusion Criteria:

* All the patients that were diagnosed as having sickle cell disease in the specific village and all the population screened for hemoglobinopathies in the same location

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients diagnosed with abnormal hemoglobin in the bedouin arab village
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Study Director — Pediatric Hematology Unit, Ha'Emek Medical Center; luci Zalman, Phd, Study Chair — Hematology Laboratory - HaEmek Medical Center; Tania Flaishman, Student, Principal Investigator — Pediatric Dpt B - Ha'Emek Medical Center
Locations (1):
- Pediatric Hematology Unit - HaEmek Medical Center, Afula, Israel